CLINICAL TRIAL: NCT06208228
Title: Effect of Kinesio-taping Technique on Oral Feeding and Swallowing Functions: An Acoustic Analysis of Swallowing Sound in Late Preterm Infants
Brief Title: Effect of Kinesio-taping Technique on Oral Feeding in Late Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Associate Proffessor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA18/36
Record Dates: First submitted 2024-01-03; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Swallow; Preterm Infant; Newborn; Kinesiotaping; Sucking
Keywords: swallow; preterm infant; newborn; kinesiotaping; sucking
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape (Experimental): Kinesiotape application to masseter and hyoid muscles of late preterm infants for improving sucking and swallowing.
  Interventions: Device: Kinesiotaping
- Control (No Intervention): In this group the late preterm infants won't be applied kinesiotaping to suck and swallow muscles.

INTERVENTIONS:
Device: Kinesiotaping — Kinesiotape application to masseter and hyoid muscles of late preterm infants for improving sucking and swallowing.
  Arms: kinesiotape

SUMMARY:
Difficulty in feeding among late preterm infants is one of the most significant factors contributing to prolonged hospitalization and re-admissions. By providing support to the sucking and swallowing muscles early in their development, the maturation process can be expedited, allowing for the safe early discharge of preterm infants.

This study aims to investigate the effects of the Kinesio taping technique on feeding muscles and assess feeding and swallowing function in late preterm infants using acoustic analysis of swallowing sounds.

DETAILED DESCRIPTION:
Problems such as poor nutrition, weak sucking, lack of suck-swallow-respiration coordination, low weight gain are among the factors increasing the risk of morbidity in late preterm infants. Early support of sucking and swallowing muscles for the development of suck-swallow coordination can shorten the maturation process and provide early discharge of late preterm infants. The aim of this study is to document kinesiotape technique to support sucking and swallowing muscles for treating nutritional problems and for reducing nutrition risks and accelerating maturation. According to power of analysis of this study, 74 infants planned to assign to kinesiotaping group or control group randomly. In kinesiotaping group, infants feeding performance will be evaluated by measuring the amount of milk invested, maximum heart rate, oxygen saturation, speed of milk intake and counting the number of swallow during feeding. Kinesiotape will be applied to masseter and hyoid muscles 24 hours later after the birth of the infant. Infants will be evaluated before kinesiotape application, 3 hour later and 24 hour later after the application.

ELIGIBILITY:
Inclusion Criteria:

* Infants born in Baskent University Ankara Hospital,
* age between 34-36.6 weeks

Exclusion Criteria:

* Infants with multiple kongenital anomaly,
* hypoxic ischemic encephalopathy,
* intraventricular and intracranial hemorrhage,
* necrotizing enterocolitis,
* tracheoesophageal fistula,
* diaphragmatic hernia,
* hydrocephalus,
* respiratory distress.

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the number of swallows of the baby during feeding | Through study completion, an average of 1 year
  digital stethoscope

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Comuk Balci, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If requested, then the investigators could share the IPD